Protocol Title: Addressing Cervical Cancer Disparity in South Florida: CBPR in Action

Version Date: 2/2/17

NCT#02202109

## Statistical Analysis

Baseline characteristics were compared across the two study arms using chi-square tests (categorical data) and t-tests (continuous data). Crude differences in proportion of women screened by study arm (overall and stratified by neighborhood site) were tested using chi-square tests. We then modeled the association between sociodemographic variables and screening completion using univariate and multivariable logistic regression analyses. We included neighborhood site, age, income, insurance status, education, Pap history, marital status and citizenship status as covariates in the multivariable analysis. Race/ethnicity was not analyzed as it was highly collinear with site (e.g. all Haitians resided in Little Haiti). We report odds ratios (ORs) and corresponding 95% confidence intervals (CI) for the regression analyses. Secondary outcomes were analyzed using paired McNemar chi-square tests for the overall sample, and stratified by neighborhood site. All statistical tests were two-sided, with significance set at the p < 0.05 level. The data were analyzed using SAS 9.4 (SAS Institute Inc., Cary, NC, USA).